CLINICAL TRIAL: NCT00558337
Title: An Efficacy, Safety, and Pharmacokinetics/Pharmacodynamic Relationship Study of L-Dopa/Carbidopa in a Novel Release Formulation in Parkinson's Disease Patients
Brief Title: Efficacy, Safety, and Pharmacokinetics/Pharmacodynamic Study of L-Dopa/Carbidopa To Treat Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Osmotica Pharmaceutical US LLC (Industry)
Responsible Party: Gustavo Fischbein, Osmotica Pharmaceutical Argentina
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: OS353-CTP 01
Record Dates: First submitted 2007-11-12; First posted 2007-11-14 (Estimated); Last update posted 2009-01-14 (Estimated); Status verified 2009-01

CONDITIONS: Parkinson's Disease
Keywords: Treatment of Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — carbidopa, levodopa drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: levodopa-carbidopa
- B (Active Comparator)
  Interventions: Drug: levodopa-carbidopa

INTERVENTIONS:
Drug: levodopa-carbidopa — novel levodopa/carbidopa formulation or a reference levodopa/carbidopa formulation

SUMMARY:
Determine if a novel levodopa/carbidopa formulation results in a better clinical response on Parkinson's Disease patients compared to the reference formulation of levodopa/carbidopa in terms of motor complications, onset of action and response duration.

DETAILED DESCRIPTION:
Primary objective is to demonstrate a better clinical response profile of novel levodopa/carbidopa formulation vs. the reference formulation of levodopa/carbidopa in patients with Parkinson's Disease as judged by motor performance and to describe pharmacokinetic profile for the novel formulation compared to the reference.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnostic of Parkinson's Disease, with a Hoehn and Yahr Staging within 2-4, and L-Dopa therapy complications
* at least 2years of L-Dopa therapy
* Patients with the ability to differentiate between "ON" and "OFF" periods
* Patients who have been receiving stable doses of L-Dopa between 600 and 1600 mg/day, for at least 2 months prior to the screening visit using a dosing regimen not higher that 5 times a day, and not expected in the investigator's opinion to need any dose modifications over the duration of the study
* Patients presenting a score of at least 2 in the UPDRS IVa, item 32 and/or a score of at least 2 in the UPDRS IVb, item 39, at screening and randomization visits based on clinical records for the first visit and daily diary cards at randomization time.
* Willing and able to understand and sign Informed Consent form

Exclusion Criteria:

* Patients with a diagnosis of any known secondary Parkinsonian syndrome, (vascular, toxin or drug-induced, metabolic or infectious, etc) or other neurodegenerative disorder with parkinsonism (Progressive Supranuclear Palsy, Corticobasal Degeneration, Multiple System Atrophy, etc).
* Patients receiving other concomitant anti-Parkinsonian pharmacological therapies affecting L-dopa or dopamine metabolisom (COMT inhibitors or MAO inhibitors)
* Subjects who have undergone prior functional neurosurgical treatment for PD (ablation or Deep Brain Stimulation).
* Patient with a L-dopa dosage regimen greater than 5 times a day which is not able to be adapted to a q.i.d. regimen.
* Patients having received L-dopa / Decarboxylase inhibitors therapy for less than 2 years.
* Patients needing nightly doses of L-dopa / Decarboxylase inhibitors apart from the four daily doses.
* Any medical condition or past medical history that, in the investigator's judgment, would increase the risk of exposure to L-dopa / Carbidopa or interfere with the evaluation of the study objectives.
* Patients with unstable or clinically significant known medical illness; such as cardiac, pulmonary, kidney, hepatic and/or gastrointestinal disease that would, in the investigator's judgment, interfere with the safe course of the study.
* Cognitive impaired patients, as determined by a score of lesser than 26 on the Mini-Mental Score Status Examination. (MMSE < 26).
* Alcohol or illegal drugs abuse.
* Pregnant or lactating patients.
* Hypersensitivity to any of the investigational drugs, based on known allergies to drugs of the same class.
* Patients having taken any research drugs over the last 30 days prior to the beginning of the study.
* Blood donation, or blood products, or participation to a clinical trial with serial blood withdrawals, within twelve weeks prior to the start of the trial, or intention to donate blood or blood products within three months following the study completion.
* Patients who have received some of the following medications with an anticipation of no more than 7 treatment-drug elimination half-lives of entry time: Dopamine D2 receptor antagonists , isoniazid, anti-epileptic drugs, IMAO A or B, pyridoxine, ferrous salts or methyldopa.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2007-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Evidence of a novel levodopa/carbidopa formulation providing a better clinical profile than reference levodopa/carbidopa formulation using Unified Parkinson's Disease Rating Scale (UPDRS III) and patient's diary cards | every half hour for the first 8 hours after dosing

SECONDARY OUTCOMES:
Other measurements to be used for demonstrating clinical profile is UPDRS II and IV, Clinical Global Impression Scale (CGI)/Patient's Global Improvement Scale (PGI), and the Abnormal Involuntary Movement Scale (AIMS) | over the course of the study

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Fischbein, M.D., Study Director — Osmotica Pharmaceutical Argentina S.A.
Locations (9):
- Argentina (9):
  - Fundacion Alfredo Thomson, Buenos Aires
  - Hospital Posadas, Buenos Aires
  - Hospital Ramos Mejía, Buenos Aires
  - Hospital Sirio Libanés, Buenos Aires
  - Instituto Frenopático, Buenos Aires
  - nstituto INEBA, Buenos Aires
  - Policlínica Bancaria, Buenos Aires
  - Fundación Rosarina de Neuro-Rehabilitación, Rosario
  - Hospital San Bernardo, Salta